CLINICAL TRIAL: NCT05821426
Title: Evaluation of the Safety and Effectiveness of Magneto eTrieve™ PE Kit for Endovascular Thrombectomy in Subjects With Acute Pulmonary Embolism
Brief Title: Evaluation of the Magneto eTrieve™ PE Kit for Endovascular Thrombectomy in Subjects With Acute Pulmonary Embolism
Acronym: eTrieve II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Magneto Thrombectomy Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KT1-CLN010
Record Dates: First submitted 2023-04-04; First posted 2023-04-20 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; eTrieve
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- eTrieve PE Kit (Experimental)
  Interventions: Device: eTrieve PE Kit

INTERVENTIONS:
Device: eTrieve PE Kit — Patients will be treated with the eTrieve PE Kit

SUMMARY:
Prospective, multi-center, open-label, single-arm clinical study of the safety and effectiveness of the eTrieve™ in subjects presenting with signs and symptoms of acute intermediate-risk pulmonary embolism

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical signs, symptoms, and presentation consistent with acute pulmonary embolism (PE)
* PE symptom duration ≤ 14 days
* Filling defect in at least one main or lobar pulmonary artery on CTA
* Right ventricle / left ventricle (RV/LV) ratio ≥ 0.9 on CTA (Investigator's reading)
* Systolic blood pressure ≥ 90 mmHg
* Stable heart rate < 130 BPM prior to the index procedure
* Anatomy that, in the opinion of the interventionalist, allows safe passage of the eTrieve™ catheters
* Written informed consent

Exclusion Criteria:

* Patients with a combined reason for their decompensation (e.g., a patient with both sepsis and PE)
* PE within 3 months prior to screening assessment
* Thrombolytic use within 30 days prior to baseline CTA
* Pulmonary hypertension with peak systolic PAP > 70 mmHg
* Inotrope or vasopressor requirement after fluid administration to keep the systolic blood pressure ≥ 90 mmHg
* Fraction of inspired Oxygen (FiO2) requirement > 40% or supplemental oxygen > 6 LPM to keep oxygen saturation > 90%
* Any of the following laboratory findings (within 6 hours prior to index procedure):

  1. Hematocrit < 28%
  2. Platelets < 100,000/µL
  3. Serum creatinine > 1.8 mg/dL
  4. INR > 3
* Major trauma Injury Severity Score (ISS) > 15 within 14 days prior to screening assessment
* Intracardiac lead in right ventricle, right atrium or coronary sinus, placed within 6 months prior to screening assessment
* Known presence of intracardiac clot
* Cardiovascular or pulmonary surgery within last 7 days
* Active malignancy and / or on chemotherapy
* Known bleeding diathesis or coagulation disorder
* Left bundle branch block
* History of severe or chronic pulmonary arterial hypertension
* History of left ventricular ejection fraction ≤ 30%
* History of decompensated heart failure
* History of underlying oxygen dependent lung disease
* History of chest irradiation
* History of Heparin Induced Thrombocytopenia (HIT)
* Any contraindication to systemic therapeutic doses of heparin or other anticoagulants
* Known anaphylactic reaction to radiographic contrast agents that cannot be adequately pre-medicated
* Known hypersensitivity or contraindication to procedural medications which cannot be adequately managed medically
* Imaging evidence or other evidence that suggests, in the opinion of the investigator, the subject is not appropriate for mechanical thrombectomy intervention
* Life expectancy of < 90 days as determined by the investigator
* Co-morbid condition(s) that, in the opinion of the investigator, could limit the patient's ability to participate in the study, including compliance with follow-up requirements, or that could impact the scientific integrity of the study
* Female who is pregnant or nursing
* Current participation in another investigational drug or device treatment study
* Previous enrollment in the eTrieve™ II Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
MAE | 48 hours
  Number of Major Adverse Event (MAE) within 48 hours post-index procedure, as adjudicated by the Clinical Events Committee (CEC)
RV/LV ratio | 48 hours
  Change in RV/LV ratio from baseline to 48 hours post-index procedure (or discharge, whichever occurs first) as assessed by the CTA core laboratory

SECONDARY OUTCOMES:
Use of thrombolytics | within 48 hours
  Use of thrombolytics within 48 hours post-index procedure
ICU/hospitalization length | within 30 days
  Length of stay in the Intensive Care Unit (ICU)/hospital, associated with the index thrombectomy procedure
Modified Miller score | at 48 hours
  Change in the Modified Miller Score between baseline and 48 hours post-index procedure as assessed by the CTA core laboratory
Mortality | within 30 days
  Mortality due to any cause within 30 days post-index procedure
Device related SAE | within 30 days
  Device-related serious adverse events within 30 days post-index procedure, as adjudicated by the CEC
PE reocurrence | within 30 days
  Symptomatic PE recurrence within 30 days post-index procedure